CLINICAL TRIAL: NCT01239459
Title: An Open-label Pharmacokinetic and Tolerability Study of Teriflunomide Given as a Single 14 mg Dose in Subjects With Severe Renal Impairment, and in Matched Subjects With Normal Renal Function
Brief Title: Pharmacokinetic and Tolerability Study of 14 mg Single Dose of Teriflunomide in Subjects With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: POP11432; 2010-022354-16 (EudraCT Number); U1111-1117-6723 (Other: UTN)
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — teriflunomide; Cholestyramine Resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe impaired renal function (Experimental): Subjects with severe renal impairment as defined by Cockroft-Gault formula
  Interventions: Drug: Teriflunomide HMR1726; Drug: Cholestyramine
- Normal renal function (Experimental): Subjects with normal renal function as defined by Cockroft-Gault formula
  Interventions: Drug: Teriflunomide HMR1726; Drug: Cholestyramine

INTERVENTIONS:
Drug: Teriflunomide HMR1726 — Pharmaceutical form:film coated tablet
  Route of administration: oral administration on Day 1 under fasted condition
Drug: Cholestyramine — Pharmaceutical form:powder
  Route of administration: oral administration 3 times per day on Day 54 and 55

SUMMARY:
Primary Objective:

- To determine the effect of severe renal impairment on the pharmacokinetic profile of teriflunomide administered as a single 14 mg dose as compared to healthy subjects

Secondary Objective:

- To assess the tolerability of teriflunomide administered as a single 14 mg dose in subjects with severe renal impairment compared to subjects with normal renal function.

DETAILED DESCRIPTION:
The total study duration per subject is 11-15 weeks broken down as follows:

* Screening: up to 3 weeks
* Hospitalization: 3 days (admission 1 day prior to study drug intake)
* Follow-up: 10 -12 weeks

ELIGIBILITY:
Inclusion criteria:

Subjects with renal impairment:

* Male subject between 18 and 75 years of age inclusive and postmenopausal female between 45 and 75 years of age inclusive.
* Chronic severe renal impairment as defined by Cockroft-Gault formula (creatinine clearance (CLcr) < 30mL/min, but not requiring hemodialysis).
* Laboratory parameters within the acceptable range for subjects with renal impairment; in particular, hepatic enzymes (ALT, AST) and bilirubin should be < 2 x upper limit of normal range and neutrophils should be within normal ranges.

Matched healthy subjects:

* Male subject between 18 and 75 years of age inclusive and postmenopausal female between 45 and 75 years of age inclusive, matched by age.
* Body weight within 15% of the body weight of the subjects with renal impairment to be matched and Body Mass Index between 18.0 and 30.0 mg/kg2 inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal renal function as defined by Cockroft-Gault formula (creatinine clearance (CLcr) > 80mL/min)
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however serum creatinine, alkaline phosphatase, hepatic enzymes (AST, ALT), bilirubin (unless the subject has documented Gilbert syndrome) should not exceed the upper limit of normal range.

Exclusion criteria:

Subjects with renal impairment:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastro-intestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female) or infectious disease, or signs of acute illness.
* Active hepatitis, hepatic insufficiency.
* Acute renal failure (de novo or superimposed to pre-existing chronic renal impairment), nephrotic syndrome.
* Subject requiring dialysis during the study.
* Any significant change in chronic treatment medication within 14-days before inclusion.
* Any drug, which could impact by any mechanism of action, the pharmacokinetic of the investigational product.
* Positive reaction to Human Immunodeficiency Virus (HIV) tests: anti-HIV1 antibodies, anti-HIV2 antibodies
* Positive results on urine drug screen (amphetamines / methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates) unless this result is secondary to a documented medical prescription.
* Positive alcohol test.
* Man who disagrees to use a double barrier method of contraception with their partner during the study.

Matched healthy subjects:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* For subjects 50 years old and below:

  * any medication (including St John's Wort) within 14 days before inclusion, or within 5 times the elimination half-life or pharmacodynamic halflife of that drug, whichever the longest, with the exception of menopausal hormone replacement therapy.
  * any significant change in chronic treatment medication within 14-days before inclusion.
* Any drug, which could impact by any mechanism of action, the pharmacokinetic of the investigational product.
* Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, antihepatitis C virus (anti-HCV) antibodies, HIV1 antibodies, anti-HIV2 antibodies.
* Positive results on urine drug screen (amphetamines / methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol test.
* Man who disagrees to use a double barrier method of contraception with their partner during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of Teriflunomide determined from plasma concentration (Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast and AUC)) | 56 days

SECONDARY OUTCOMES:
Clinical safety evaluation (AE reporting, laboratory tests (hematology, biochemistry and urinalysis), vital signs and ECG parameters) | Up to 12 weeks (until the end of study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Berlin, Germany